CLINICAL TRIAL: NCT03303833
Title: The GEOLynch Cohort Study: Genetic, Environmental and Other Factors That Influence Tumour Risk Among Persons With Lynch Syndrome
Brief Title: The GEOLynch Cohort Study
Acronym: GEOLynch
Status: Recruiting | Type: Observational
Sponsor: Wageningen University (Other)
Collaborators: Wereld Kanker Onderzoek Fonds (Other); Dutch Cancer Society (Other); Funding: Biobanking and BioMolecular resources Research Infrastructure The Netherlands (Unknown)
Responsible Party: Sponsor
Other Study IDs: CMO 2005-283; 2014/1184 (Other Grant/Funding Number: Wereld Kanker Onderzoek Fonds (WCRF NL)); 2005-3275 / 2007-3842 (Other Grant/Funding Number: Dutch Cancer Society (KWF)); CP2013-58 (Other Grant/Funding Number: Biobanking and BioMolecular resources Research Infrastructure The Netherlands (BBMRI))
Record Dates: First submitted 2017-09-14; First posted 2017-10-06 (Actual); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Lynch Syndrome; Neoplasms; Hereditary Nonpolyposis Colorectal Cancer; Colorectal Neoplasms
Keywords: Lifestyle; Nutrition
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis; Neoplasms; Colorectal Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Buccal swabs and blood samples.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Persons with Lynch syndrome
  Interventions: Other: No intervention, observational study.

INTERVENTIONS:
Other: No intervention, observational study.

SUMMARY:
The GEOLynch cohort study has been established to investigate the influence of genetic, environmental and other factors on tumour risk in persons with Lynch syndrome.

DETAILED DESCRIPTION:
The GEOLynch cohort study includes persons with Lynch syndrome (LS) only. Persons with LS carry an inherited mutation in one of the DNA mismatch repair genes MLH1, MSH2, MSH6 or PMS2 which increases their risk of several types of cancer, especially colorectal and endometrial cancer. Additionally, mutations in the EPCAM gene that result in epigenetic silencing of the MSH2 gene cause LS. Since 2006, persons with LS are invited to participate in the GEOLynch cohort study via the Netherlands Foundation for the Detection of Hereditary Tumours, the Radboud University Medical Center Nijmegen or the University Medical Centre Groningen. Moreover, persons with LS can participate in the study after contacting the researcher themselves. Participants are asked to complete a food frequency questionnaire and questionnaires about dietary supplement use, physical activity, weight, height and medication use. A buccal swab was asked of every participant recruited between 2006 and 2008. From 2012 on, newly recruited participants are asked to donate a blood sample instead of a buccal swab. Furthermore, participants who had been recruited between 2006 and 2008 were asked to complete the questionnaires again and to donate a blood sample too. Hence, follow-up measurements are available for a subset of participants. DNA has been subtracted from the buccal swabs to genotype SNPs of the IGF gene axis and polymorphisms of MTHFR C377T. Blood samples are biobanked to facilitate future analyses of biomarkers, nutrients, DNA etc. Clinical characteristics regarding performed colonoscopies and tumour diagnoses of all participants is gathered from medical records and a linkage to the nationwide network and registry of histo- and cytopathology in the Netherlands (PALGA Foundation ). Hazard ratios will be calculated to investigate the influence of genetic, environmental and other factor on tumour risk. Repeated measures analyses will be used if follow-up measurements are taken into account.

ELIGIBILITY:
Inclusion Criteria:

* Persons with a known mutation in a gene that causes Lynch syndrome, i.e. with an inherited monoallelic pathogenic germline mutation in either the MLH1, MSH2, MSH6, PMS2 or EPCAM gene.
* Aged between 18 and 80 years at inclusion.

Exclusion Criteria:

* Additional carrier of another hereditary colon cancer predisposition syndrome (e.g. FAP)
* (Chronic) Inflammatory bowel disease
* Non-Dutch speaking
* Dementia or another mental condition that makes it impossible to fill out questionnaires
* Terminally ill persons

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women aged 18 to 80 years with Lynch syndrome who do or do not have a (previous) cancer diagnosis.
Enrollment: 1000 (Estimated)
Dates: Start 2006-07-01 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Colorectal tumour diagnoses | Diagnoses before and after study inclusion will be assessed approximately every 2 years until study completion by regularly reviewing medical reports and/or pathology reports.
  All diagnosed colorectal adenomas and carcinomas described in paticipants' medical reports and/or pathology reports.
Endometrial cancer diagnoses | Diagnoses before and after study inclusion will be assessed approximately every 2 years until study completion by regularly reviewing medical reports and/or pathology reports.
  All diagnosed endometrial cancers described in participants' medical reports and/or pathology reports.
Overall cancer diagnoses | Diagnoses before and after study inclusion will be assessed approximately every 2 years until study completion by regularly reviewing medical reports and/or pathology reports.
  All diagnosed cancer types described in participants' medical reports and/or pathology reports.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Kampman, PhD, Principal Investigator — Wageningen University
Locations (1):
- Wageningen University, Wageningen, Netherlands

REFERENCES:
- [Background] van Duijnhoven FJ, Botma A, Winkels R, Nagengast FM, Vasen HF, Kampman E. Do lifestyle factors influence colorectal cancer risk in Lynch syndrome? Fam Cancer. 2013 Jun;12(2):285-93. doi: 10.1007/s10689-013-9645-8. PMID 23657759
- [Result] Jung AY, van Duijnhoven FJ, Nagengast FM, Botma A, Heine-Broring RC, Kleibeuker JH, Vasen HF, Harryvan JL, Winkels RM, Kampman E. Dietary B vitamin and methionine intake and MTHFR C677T genotype on risk of colorectal tumors in Lynch syndrome: the GEOLynch cohort study. Cancer Causes Control. 2014 Sep;25(9):1119-29. doi: 10.1007/s10552-014-0412-4. Epub 2014 Jun 12. PMID 24916333
- [Result] Botma A, Nagengast FM, Braem MG, Hendriks JC, Kleibeuker JH, Vasen HF, Kampman E. Body mass index increases risk of colorectal adenomas in men with Lynch syndrome: the GEOLynch cohort study. J Clin Oncol. 2010 Oct 1;28(28):4346-53. doi: 10.1200/JCO.2010.28.0453. Epub 2010 Aug 23. PMID 20733131
- [Result] Winkels RM, Botma A, Van Duijnhoven FJ, Nagengast FM, Kleibeuker JH, Vasen HF, Kampman E. Smoking increases the risk for colorectal adenomas in patients with Lynch syndrome. Gastroenterology. 2012 Feb;142(2):241-7. doi: 10.1053/j.gastro.2011.10.033. Epub 2011 Nov 4. PMID 22062356
- [Result] Botma A, Vasen HF, van Duijnhoven FJ, Kleibeuker JH, Nagengast FM, Kampman E. Dietary patterns and colorectal adenomas in Lynch syndrome: the GEOLynch cohort study. Cancer. 2013 Feb 1;119(3):512-21. doi: 10.1002/cncr.27726. Epub 2012 Dec 17. PMID 23254892
- [Result] Heine-Broring RC, Winkels RM, Botma A, van Duijnhoven FJ, Jung AY, Kleibeuker JH, Nagengast FM, Vasen HF, Kampman E. Dietary Supplement Use and Colorectal Adenoma Risk in Individuals with Lynch Syndrome: The GEOLynch Cohort Study. PLoS One. 2013 Jun 18;8(6):e66819. doi: 10.1371/journal.pone.0066819. Print 2013. PMID 23825568
- See also: GEOLynch website — http://www.geolynch-studie.nl/geolynchstudy_eng